CLINICAL TRIAL: NCT03167060
Title: Nasal Cavity Cooling for the Symptomatic Relief of Migraine Headache - A Randomized, Double Blind, Placebo Controlled Study" , the BrainCool-Migraine Study
Brief Title: BrainCool-Migraine Intranasal Cooling Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumbria Partnership NHS Foundation Trust (Other)
Collaborators: BrainCool AB (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CP1628
Record Dates: First submitted 2017-05-19; First posted 2017-05-25 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: Post-market clinical study of one or more CE marked devices within intended purposes, involving a change to standard care or randomisation between groups
Who Masked: Participant
Masking Description: Controls will undergo same treatment with the medical device, but it will be a sham treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Rhinochill (Active Comparator): Intranasal cooling device , using nasal cannula
  Interventions: Device: Active RhinoChill
- Control Rhinochill (Sham Comparator): Intranasal cooling device , using nasal cannula (difference with active device not disclosed to maintain blindness)
  Interventions: Device: Control Rhinochill

INTERVENTIONS:
Device: Active RhinoChill — Participants will be provided with a RhinoChill® device (Active) and an Intranasal Migraine catheter. Once they have the RhinoChill® device, they are asked to treat the next two of your migraines with the device. This requires a maximum of 10 minute intra-nasal treatment as soon as possible after the start of your migraine.
  The participation in the trial will last until 3 migraine headaches have been treated with the RhinoChill® device.
  Arms: Active Rhinochill
Device: Control Rhinochill — Participants will be provided with a RhinoChill® device (Sham) and an Intranasal Migraine catheter. Once they have the RhinoChill® device, they are asked to treat the next two of your migraines with the device. This requires a maximum of 10 minute intra-nasal treatment as soon as possible after the start of your migraine.
  The participation in the trial will last until 3 migraine headaches have been treated with the RhinoChill® device.
  Arms: Control Rhinochill

SUMMARY:
This study will be a randomised placebo controlled trial examining the effectiveness of using an intranasal evaporative cooling device (the RhinoChill intransal device) in providing relief of pain and symptoms of acute migraine.The treatment works by introducing cooling into the passageways of the nose through two small cannulas thereby cooling the local nasal tissue and the blood vessels which supply blood to the brain. This cooling effect will cause the blood vessels to constrict as well as stimulating special cold receptors that are thought to be involved in the relief of migraine, thereby providing both pain and associated symptomatic relief. In total, 90 patients randomised in a 1:1 fashio n will be recruited from three different NHS Trusts. The patients will have a 30-day period of data collection for their current migraine frequency, treatment and response to medication (with a minimum of 2 migraine attacks recorded) before starting the treatment phase with the RhinoChill Device. Treatment will be for 3 migraine attacks. Only a single treatment is allowed for the first attack, but on the second attack the patient may deliver 2 treatments with a gap of at least 2 hours between treatments, if indicated.

DETAILED DESCRIPTION:
Mechanical techniques to alleviate migraine symptoms have been used for many years, cooling and compression being the most frequently applied. Cryotherapy is the most common non-pharmacological self-administered pain-relieving method currently used by migraine sufferers. The first manuscript documenting the application of ice mixtures was published by James Arnott in 1849. Simple techniques based on cryotherapy, using various methods of cold and ice application have been reported over the last three decades. Friedman described a device using hollow metal tubes cooled by circulating cold water, applied to the periapical area of the maxillary molars. Sprouse-Blum reported benefit from applying frozen icepacks targeting carotid arteries at the front of the neck in migraine treatment.

Several pathophysiological mechanisms of action have been proposed. These mechanisms include:

1. Neurovascular mechanism: Application of cold induces vasoconstriction with subsequent decreased downstream blood flow. This leads to inhibition of the release of inflammatory mediators which results in decreased vascular permeability and local oedema.
2. Pain gating by differential effect on nerve conduction: Cryotherapy induces analgesia by slowing nerve conduction velocity, with small myelinated fibers being affected first, followed by large myelinated fibers and the unmyelinated fibers being affected last. Via mechanism of the gate control of pain, affecting the small myelinated nociceptive pain afferents first, cryotherapy induces analgesia.
3. Metabolic mechanism: Cryotherapy decreases metabolic and enzymatic activity, due to reduced demand for adenosine triphosphate (ATP) and oxygen.
4. Transient Receptor Potential (TRP) channels: Recent studies suggest that TRP channels may have a role in headache and pain genesis due to their response to environmental stimuli such as temperature changes.

The nasal cavity provides a large diffuse surface area that is highly vascular. Cooling via the nasal cavity therefore offers the ability to cool across the thin cribriform plate via both direct conductive mechanisms that do not rely on spontaneous circulation as well as indirect haematogenous mechanisms. Numerous subarachnoid and pial arterial branches exposed to the cerebrospinal fluid (CSF) have diameters in the range of the vessels of the retia mirabilia of animals in which selective brain cooling has been clearly established experimentally. Vascular anatomy allows transfer of venous blood from the skin of the head as well as nasal and paranasal mucous membranes to the dura mater thereby providing an excellent basis for the convective process of intranasal evaporative cooling. The dura mater, with its high vascularization, may transmit temperature changes to the CSF compartment, which may influence the temperature of brain parenchyma directly or indirectly, via brain arteries.

We suppose that another effect of intranasal cooling may be local vasoconstriction and subsequent associated vasoconstriction of cerebral arteries due to the presence of the nebulized coolant in the nasal cavity.

Many sufferers use mechanical techniques to relieve the headache. Simple techniques that have been recommended and tried include cryotherapy. Applying an icepack to the painful area has been the most frequently mentioned method. Many studies demonstrating the effectiveness of a variety of non-pharmacological modalities have been reviewed over the years. Although definite proof of effectiveness through traditional scientific method has been lacking in most instances. There is a trial reported by Friedman, where intraoral cooling was applied. Significant migraine relief has been obtained from chilling confined to the area. Thirty-five symptomatic episodic migraine patients were enrolled in this study, comparing 40 minutes of bilateral intraoral chilling, 50 mg of oral sumatriptan, and 40 minutes of sham (tongue) chilling. Hollow metal tubes chilled by circulating ice water were held in the maxillary molar periapical areas by the patient. Pain and nausea were recorded at baseline and 1, 2, 4, and 24 hours after start of treatment, using a numeric symptom-relief scale. Significant mean headache relief was obtained by maxillary chilling and sumatriptan at all four time intervals, with poor relief obtained by placebo. Maxillary chilling was more effective than sumatriptan at all four time intervals. Significant nausea relief was obtained by maxillary chilling and sumatriptan at post treatment and 2 and 4 hours later. At 24 hours, some headache and nausea recurrence was noted with sumatriptan. The repeated-measures analysis of variance indicated that both treatments, drug (P = 0.024) and maxillary chilling (P = 0.001), reduced the headache, as compared with the control group. Tenderness in the premolar area suggests local inflammation associated with vasodilatation and oedema. Because chilling can resolve local oedema, authors raised the possibility that an intraoral inflammation may be a factor in migraine aetiology. Although it is a possibility the cooling effect might have caused indirect vasoconstriction of the dilated meningeal blood vessels.

In the COOLHEAD 1 trial, investigators found that the use of RhinoChill® intranasal cooling within a clinic environment for 15 patients provided a statistically significant reduction of pain and associated symptoms of migraine at 5 minutes and 10 minutes (during treatment), and at 1 hour and 2 hours following treatment (all p values <0.001) along with a significant effect on pain and symptoms at 24 hours (p <0.001). In total, 87% of patients enrolled into the trial received a treatment benefit following from a short term (<20minutes) period of intranasal cooling.

Enrollment into the trial was challenging as participants were required to present at the hospital clinic for treatment between the hours of 9am to 7pm Monday to Friday, which for some, was too difficult while undergoing a migraine headache, and for others, the centre was not open for treatment at the time of their migraines. For those that did come in for treatment, it was found to be burdensome to travel while a migraine was present.

The results of this trial demonstrate that the RhinoChill® intranasal cooling device is both safe and effective to treat migraine patients within the setting of a hospital clinic environment. In this planned BrainCool-Migraine trial, the treatment will be self-administered by the patient. To allow for a swifter enrollment of patients into the study, to evaluate this treatment methodology in an as close to real world environment as possible, and to minimize any burden or discomfort to the patient by traveling to the hospital clinic with an active migraine headache on the one hand and to achieve best possible control of the study on the other hand, the self-administration by the patient in this study will be allowed and required to be done at home, as opposed to the clinic or any other location. The proven treatment methods and procedures as examined and described in the COOLHEAD 1 in-clinic trial will be implemented throughout the BrainCool-Migraine trial treatment procedures so as to ensure the high quality and standards associated with the previous trial.

It is recognised that migraine treatments are prone to placebo effects, which is further enhanced by the use of a medical device in an in-hospital setting, therefore in this BrainCool-Migraine trial, the design will be that of a double blinded, randomised, two arm, placebo control multicentre clinical trial.

The hypothesis we propose is that the application of RhinoChill® nasal cavity cooling will provide effective relief of pain and symptoms associated with episodic migraine (with or without aura). The null hypothesis is that no significant difference in pain scores, headache response or symptom severity scores will be found between the active treatment and placebo groups.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years old or over and ≤70 years of age.
* Migraine diagnosis of at least 1 year
* Migraine attacks between 1 and 15 per month
* Onset of first migraine < 50 years of age
* Migraine prophylaxis medication unchanged for 3 months prior to enrollment
* Meets International Classification for Headache Disorders (2nd Edition) criteria for diagnosis of Episodic Migraine with or without aura
* Able to attend a short training session on the practical use of the RhinoChill® device and agrees to only use the device as instructed and as laid out in the official instructions for use

Exclusion Criteria:

* < 18 and >70 years of age
* Known oxygen dependency to maintain SaO2 >95%
* Diagnosed Hypertensive and currently uncontrolled with Systolic BP > 140mmHg and Diastolic BP > 90mmHg on baseline assessment.
* Marked nasal septal deviation, recurrent epistaxis or chronic Rhino-Sinusitis.
* Intranasal obstruction preventing full insertion of nasal catheter.
* Known base of skull fracture or facial trauma
* Concurrent sinus/intranasal surgery
* Diagnosed with Thromobocytopenia
* Previous Stroke or Myocardial Infarction
* Unable to fully understand the consent process and provide informed consent due to either language barriers or mental capacity
* Previously enrolled into the COOLHEAD 1 trial.
* No recorded migraine following initial 30 day data collection period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-02-06 (Actual)

PRIMARY OUTCOMES:
Participant is pain free at two hours following trial device treatment The patients' first treatment will be used for analysis of the superiority of the rate of patients pain free at two hours following treatment for those receiving the standard R | two hours
  The first treatment with the RhinoChill device will be used for analysis of the superiority of the rate of participants who are pain free at two hours following treatment for those receiving the standard RhinoChill® treatment. This will be compared to those participants who are randomised to receive sham device treatment. Likert scale questionnaire will record the outcome

SECONDARY OUTCOMES:
Percentage of patients pain free immediately after treatment (10 minutes), at 1 hour, and 24 hours following treatment | 10 minutes, 1 hour, 24 hours
  Likert scale questionnaire will record the outcome
Headache response | 10 min, 1 hour, 2 hours, 24 hours
  Improvement of pain from severe/moderate to mild/none immediately following treatment (10 minutes), at 1 hour, 2 hours, and 24 hours following treatment. Likert scale questionnaire will record the outcome
relapse incidence | 2 hours, 48 hours
  frequency of headache return between 2 and 48 hours after the intervention. Binary outcome questionnaire
Sustained pain freedom | 2 hours, 48 hours
  pain free at 2 hours with no use of rescue medication or relapse within toal of 48 hours after treatment commenced. Likert scale questionnaire will record the outcome
Total migraine freedom | 2 hours
  absence of pain, nausea, photophobia and phonophobia at 2 hours. Likert scale questionnaire will record the outcome

CONTACTS AND LOCATIONS:
Overall Officials: Jitka Vanderpol, MD, Principal Investigator — Cumbria Partnership NHS Foundation Trust
Locations (4):
- United Kingdom (4):
  - Neurosciences department, Penrith Hospital, Cumbria Partnership NHS Foundation Trust, Penrith, Cumbria
  - South tees Hospital, Middlesbrough
  - The Newcastle upon Tyne Hospitals, Newcastle upon Tyne
  - City Hospital, Sunderland, UK, Sunderland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friedman MH, Peterson SJ, Behar CF, Zaidi Z. Intraoral chilling versus oral sumatriptan for acute migraine. Heart Dis. 2001 Nov-Dec;3(6):357-61. doi: 10.1097/00132580-200111000-00003. PMID 11975819
- [Background] Sprouse-Blum AS, Gabriel AK, Brown JP, Yee MH. Randomized controlled trial: targeted neck cooling in the treatment of the migraine patient. Hawaii J Med Public Health. 2013 Jul;72(7):237-41. PMID 23901394
- [Background] Vanderpol J, Bishop B, Matharu M, Glencorse M. Therapeutic effect of intranasal evaporative cooling in patients with migraine: a pilot study. J Headache Pain. 2015 Jan 26;16:5. doi: 10.1186/1129-2377-16-5. PMID 25623151
- [Background] Zanchin G, Maggioni F, Granella F, Rossi P, Falco L, Manzoni GC. Self-administered pain-relieving manoeuvres in primary headaches. Cephalalgia. 2001 Sep;21(7):718-26. doi: 10.1046/j.1468-2982.2001.00199.x. PMID 11594999
- [Background] Diamond S, Freitag FG. Cold as an adjunctive therapy for headache. Postgrad Med. 1986 Jan;79(1):305-9. doi: 10.1080/00325481.1986.11699255. PMID 3941818